CLINICAL TRIAL: NCT05525026
Title: Evaluation of Safety and Efficacy of the BTL-785F Device for Non-invasive Facial Remodeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS500
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Non-invasive facial remodeling (Experimental): Treatment with the BTL-785-7 applicator to the BTL-785F system.
  Interventions: Device: BTL-785-7

INTERVENTIONS:
Device: BTL-785-7 — Treatment with the BTL-785-7 applicator to the BTL-785F system.

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-785F system equipped with the BTL-785-7 applicator for non-invasive facial remodeling.

DETAILED DESCRIPTION:
The study is a multicenter single-arm, open-label, interventional study. The subjects will be enrolled and assigned into a single experimental study arm. The subjects will be required to complete four (4) treatment visits and two follow-up visits.

At the baseline visit health status will be assessed and, if needed, additional tests will be performed. Inclusion and exclusion criteria will be verified and informed consent will be signed.

The treatment administration phase consists of four (4) treatment visits, delivered 5-10 days apart.

Safety measures will include documentation of adverse events (AE) including the subject's experience of pain or discomfort after the procedure. Occurrence of AE's will be checked immediately after the first treatment visit, prior/post to every other procedure and at the follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment for facial remodeling
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible sagging skin in the treated area when the face is relaxed as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Local bacterial or viral infection in the area to be treated
* Local acute inflammation in the area to be treated
* Isotretinoin and tretinoin-containing medication use in the past 12 months
* Impaired immune system caused by any immunosuppressive illness, disease or medication
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants1
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of skin disorders, keloids, abnormal wound healing and dry or fragile skin
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Nerve insensitivity (sensitivity disorders) to heat in the treatment area
* Varicose veins, pronounced edemas
* Prior use of dermal fillers, botulinum toxin, lasers, etc. therapies in the treated area that can influence the study results at the investigator discretion
* Unwillingness/inability to not change their usual cosmetics and especially not to use anti-aging or facelift products in the treated area during the duration of the study including the follow-up period
* Electroanalgesia without exact diagnosis of pain etiology
* Neurological disorders (such as multiple cerebrospinal sclerosis, epilepsy)
* Blood vessels and lymphatic vessels inflammation
* Any other disease or condition (e.g. eye disease) at the investigator discretion that may pose risk to the patient or compromise the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Non-invasive facial remodeling | 5 months
  Evaluation of facial skin appearance based on photographs before and after the study procedure according to the Global Aesthetic Improvement Scale.The GAIS is a clinically validated assessment tool used to assess overall aesthetic improvement such as facelift on a scale from -1 through 3, where the higher score is considered better.

SECONDARY OUTCOMES:
Evaluation of skin quality and aesthetic change of the treated areas after the therapies | 5 months
  Evaluation of skin quality and aesthetic change of the treated areas after the therapies based on photographs before and after the study procedure according to the Global Aesthetic Improvement Scale. The GAIS is a clinically validated assessment tool used to assess overall aesthetic improvement such as facelift on a scale from -1 through 3, where the higher score is considered better.
Subject Satisfaction | 5 months
  The Subject Satisfaction questionnaire will be used for evaluating the satisfaction. The Subject Satisfaction Questionnaire will be given to subjects after the last treatment, at 1-month and 3-month follow-up. The answers to the questions related to the subjects' overall skin and face appearance will vary from "strongly agree" to "strongly disagree".
Therapy Comfort | 5 months
  The 5-point Likert scale Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. Pain sensation will be rated by the subjects from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dr Bryan Kinney, Beverly Hills, California
  - BOYD Beauty, Birmingham, Michigan

IPD SHARING:
Plan to Share IPD: No